CLINICAL TRIAL: NCT06440967
Title: A Randomized, Placebo-controlled, Double-blind, Phase 3 Clinical Study to Investigate the Efficacy and Safety of Fezolinetant for Treatment of Moderate to Severe Vasomotor Symptoms (Hot Flashes) in Women With Stage 0 to 3 Hormone Receptor-positive Breast Cancer Who Are Receiving Adjuvant Endocrine Therapy
Brief Title: A Study to Confirm if Fezolinetant Helps Reduce Hot Flashes in Women With Breast Cancer Who Are Having Hormone Therapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2693-CL-1303; 2024-510719-31-00 (Other: CTIS (EU))
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Hot Flashes
Keywords: ESN364;; vasomotor symptoms;; fezolinetant;; VEOZAH™
MeSH Terms: conditions — Hot Flashes | interventions — fezolinetant; Tamoxifen; Aromatase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fezolinetant (Experimental): Participants taking tamoxifen or an aromatase inhibitor will receive fezolinetant once daily for 52 weeks. After the end of the 52 week treatment period, participants will continue to participate in the extension follow up until week 104. They will continue to receive the adjuvant endocrine therapy as needed.
  Interventions: Drug: Fezolinetant; Drug: Tamoxifen; Drug: Aromatase inhibitor
- Placebo (Placebo Comparator): Participants taking tamoxifen or an aromatase inhibitor will receive matching placebo once daily for 52 weeks. After the end of the 52 week treatment period, participants will continue to participate in the extension follow up until week 104. They will continue to receive the adjuvant endocrine therapy as needed.
  Interventions: Drug: Placebo; Drug: Tamoxifen; Drug: Aromatase inhibitor

INTERVENTIONS:
Drug: Fezolinetant — oral
  Other Names: ESN364;; VEOZAH™
  Arms: Fezolinetant
Drug: Placebo — oral
  Arms: Placebo
Drug: Tamoxifen — oral
Drug: Aromatase inhibitor — oral

SUMMARY:
One of the standard treatments for women with breast cancer is hormone therapy, but this treatment can cause hot flashes. Hormone replacement therapy, or HRT, is most often prescribed for hot flashes for women in menopause but cannot be given to women on hormone therapy for breast cancer. Fezolinetant, an alternative to HRT, treats hot flashes for women in menopause. As hot flashes happen in the same way for women on hormone therapy for breast cancer, fezolinetant could help these women. In this study, women on hormone therapy for breast cancer who have moderate to severe hot flashes will take part. They will either take fezolinetant or a placebo to treat their hot flashes. The placebo looks like fezolinetant but doesn't have any medicine in it.

The main aim of this study is to confirm if women who take fezolinetant have fewer hot flashes that are less severe compared to women who take the placebo.

Women 18 years or older seeking treatment for hot flashes. They can take part in the study if they have an average of 7 or more moderate to severe hot flashes each day. They are having hormone therapy for breast cancer from stage 0 (cancer cells that have not spread to nearby tissue) up to stage 3+ (the cancer has spread from the breast to the lymph nodes near the breast or the chest wall).

The women will be assigned 1 of 2 study treatments (fezolinetant or placebo) by chance alone. Treatment will be double-blinded. That means that the women in the study and the study doctors will not know who takes which of the study treatments (fezolinetant or placebo). Women who take part in the study will take 1 tablet every day for 52 weeks (1 year). Each woman will be given an electronic handheld device with an app to track their hot flashes on a daily basis. Some women may be able to use the app on their own smartphone. They will also use another device to answer questions about how hot flashes affect their daily life. During the study, the women will visit their study clinic about every 4 weeks for a health check. The last clinic visit will be 3 weeks after the women take their last tablet of study treatment (fezolinetant or placebo). After this visit the women will be called twice to check their health. The women will be in the study for about 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a personal history of stage 0-3 hormone receptor positive (HR+), either human epidermal growth factor receptor (HER)-2+ or HER-2- breast cancer; appropriate documentation includes a written or electronic report.
* Participant must be receiving stable maintenance adjuvant endocrine therapy (e.g., tamoxifen or aromatase inhibitors, such as anastrozole, letrozole and exemestane) with or without gonadotropin-releasing hormone (GnRH) agonists/antagonists for a minimum of 4 months prior to randomization and be planning to continue on adjuvant endocrine therapy for the duration of the trial without change to therapy, brand or dose. If the participant is taking GnRH agonists/antagonists, therapy must also be stable for a minimum of 4 months prior to randomization. Add-on therapies for breast cancer adjuvant treatment (e.g., cyclin dependent kinase-4 (CDK4) inhibitors) are allowed.
* Participant has a minimum average of 7 moderate to severe hot flashes (HFs) (vasomotor symptoms (VMS)) per day as recorded in the electronic daily diary (data must be available for at least 7 of the last 10 days prior to randomization).
* Has an European Cooperative Oncology Group (ECOG) score 0 or 1.
* Has at least 12-month life expectation.
* Participant is born female.
* Female participant: Is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who has a negative urine or serum pregnancy test at screening and day 1 and agrees to follow the contraceptive guidance from the time of informed consent through at least 30 days after final investigational study intervention administration.
* Female participant: Must not be breastfeeding or lactating starting at screening and while the participant is taking investigational study intervention and for 30 days after final investigational study intervention administration.
* Female participant: Must not donate ova starting at first administration of study intervention and while the participant is taking investigational study intervention and for 30 days after final investigational study intervention administration.
* Participant agrees not to participate in another interventional study while participating in the present study until the end of the 1-year extension follow-up period.
* Participant's condition is stable as determined on the basis of medical history and general physical examination, hematology and biochemistry parameters, pulse rate and/or blood pressure and electrocardiogram (ECG) (or showing no clinically relevant deviations obtained within the last 3 months or at screening).
* Participant has no new clinically significant findings on breast examination or from imaging (mammogram, breast ultrasound or equivalent). Results indicate that the participant is a good candidate for the study. Appropriate documentation includes a written or electronic report. In case of double mastectomy, imaging is not needed.
* Participant has a negative serology panel (including hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody and human immunodeficiency virus (HIV) antibody screens).

Exclusion Criteria:

* Participant has diagnosis of metastatic breast cancer (stage 4).
* Participant has current or history (except complete remission for 5 years or more prior to signing informed consent) of any malignancy except for HR+ breast cancer (stage 0 to 3) or basal cell carcinoma.
* Participant has had surgery or non-surgical (chemotherapy or radiotherapy) treatment for breast cancer within the last 3 months prior to signing informed consent.
* Participant has active liver disease, jaundice, or elevated liver aminotransferases (alanine aminotransferase (ALT) or aspartate aminotransferase (AST)), elevated total bilirubin (TBL) or direct bilirubin (DBL), or elevated alkaline phosphatase (ALP) at screening. A participant with mildly elevated ALT or AST up to < 2 × upper limit of normal (ULN) can be enrolled if TBL and DBL are normal. Participant with mildly elevated ALP (up to < 1.5 × ULN) can be enrolled if cholestatic liver disease is excluded and no cause other than fatty liver is diagnosed. Participant with Gilbert's syndrome with elevated TBL may be enrolled as long as DBL, hemoglobin and reticulocytes are normal.
* Participant has creatinine > 1.5 x ULN; or estimated glomerular filtration rate (eGFR) using the Modification of Diet in Renal Disease formula < 30 mL/min/1.73 m2 at the screening visit.
* Participant has a history of endometrial hyperplasia (participant can be enrolled if she has undergone a hysterectomy) or uterine/endometrial cancer.
* Participant has a medical condition or chronic disease (including history of neurological [including cognitive], hepatic, renal, cardiovascular, gastrointestinal, pulmonary [e.g., moderate asthma], endocrine, or gynecological disease) or malignancy that could confound interpretation of the study outcome.
* Participant uses a prohibited therapy (menopause hormone therapy (MHT), estradiol-containing hormonal contraceptive progestin and progesterone-only medicines, any treatment for VMS [prescription medications, over-the-counter, or herbal] or CYP1A2 (cytochrome P450) inhibitors) or is not willing to wash out such drugs; in addition, medications that are contraindicated due to underlying breast cancer diagnosis and the adjuvant endocrine therapy.
* Participant has a known substance abuse or alcohol addiction within 6 months of screening.
* Participant has received any investigational therapy within 90 days or 5 half-lives, whichever is longer, prior to screening.
* Participant has any condition, which makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to fezolinetant, the adjuvant endocrine therapy being used, or any components of the formulations used.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean change from Baseline to Week 4 in the frequency of moderate to severe VMS | Baseline to Week 4
  Frequency of moderate and severe vasomotor symptoms (VMS) events will be calculated as the sum of moderate and severe VMS events per day.
Mean change from Baseline to Week 12 in the frequency of moderate to severe VMS | Baseline to Week 12
  Frequency of moderate and severe VMS events will be calculated as the sum of moderate and severe VMS events per day.
Mean change from Baseline to Week 4 in the severity of moderate to severe VMS | Baseline to Week 4
  The severity of VMS will be calculated using a weighted average of VMS events.
Mean change from Baseline to Week 12 in the severity of moderate to severe VMS | Baseline to Week 12
  The severity of VMS will be calculated using a weighted average of VMS events.

SECONDARY OUTCOMES:
Mean change from Baseline to Week 12 in the MENQOL VMS 1 week recall domain score | Baseline to Week 12
  The Menopause-specific Quality of Life Questionnaire (MENQOL) is a 29-item patient-reported outcome (PRO) measure that assesses the impact of 4 domains of menopausal symptoms, as experienced over the last week: vasomotor, psychosocial, physical and sexual. Each item score ranges from 1 to 8, and each domain is scored separately; each domain mean ranges from 1 to 8. The overall questionnaire score is the mean of the domain means. Higher scores represent more bothersome menopausal symptoms. A reduction (improvement) of 1 is the minimum clinically important difference in MENQoL.
Mean Change from Baseline to Week 12 in the PROMIS SD SF 8b Total (raw) Score | Baseline to Week 12
  The Patient-reported Outcomes Measurement Information System Sleep Disturbance - Short Form 8b (PROMIS SD SF 8b) assesses self-reported sleep disturbance over the past 7 days and includes perceptions of: restless sleep; satisfaction with sleep; refreshing sleep; difficulties sleeping, getting to sleep or staying asleep; amount of sleep; and sleep quality. Responses to each of the 8 items range from 1 to 5 and the range of possible summed raw scores is 8 to 40. Higher scores on the PROMIS SD SF 8b indicate more of the concept measured (disturbed sleep).
Mean change from Baseline to Week 24 in the frequency of moderate to severe VMS | Baseline to Week 24
  Frequency of moderate and severe VMS events will be calculated as the sum of moderate and severe VMS events per day.
Mean Change from Baseline to Week 24 in the severity of moderate to severe VMS | Baseline to Week 24
  The severity of VMS will be calculated using a weighted average of VMS events.
Number of participants with Treatment Emergent Adverse Events (TEAEs) | Up to Week 55
  A TEAE is defined as Adverse Event (AE) observed after starting administration of the investigational study intervention and up to 21 days after the last dose of investigational study intervention.
Number of participants with Adverse Events of Special Interest (AESIs) | Up to Week 55
  AEs of special interest in this study will include: Progression of breast cancer including metastasis; Adverse events of uterine bleeding; Adverse events of liver test elevations; Any liver AE leading to discontinuation.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to Week 55
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or adverse events (AEs) | Up to Week 55
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) | Up to Week 52
  Number of participants with potentially clinically significant ECG values.
Mean change from Baseline in the frequency of moderate to severe VMS to the average frequency of moderate to severe VMS over Weeks 1 to 3 | Baseline and Weeks 1 to 3
  Frequency of moderate and severe VMS events will be calculated as the sum of moderate and severe VMS events per day.
Mean Change from Baseline in the frequency of moderate to severe VMS to the average frequency of moderate to severe VMS over Weeks 5 to 11 | Baseline and Weeks 5 to 11
  Frequency of moderate and severe VMS events will be calculated as the sum of moderate and severe VMS events per day.
Mean change from Baseline in the severity of moderate to severe VMS to the average severity of moderate to severe VMS over weeks 1 to 3 | Baseline and Weeks 1 to 3
  The severity of VMS will be calculated using a weighted average of VMS events.
Mean Change from Baseline in the severity of moderate to severe VMS to the average severity of moderate to severe VMS over weeks 5 to 11 | Baseline and Weeks 5 to 11
  The severity of VMS will be calculated using a weighted average of VMS events.
Percent reduction >/= 50% in the frequency of moderate and severe VMS from baseline | Baseline to Weeks 1, 4, 8 and 12
  Frequency of moderate and severe VMS events will be calculated as the sum of moderate and severe VMS events per day. Percent reduction of >/= 50% will be reported.
Percent reduction >/= 75% in the frequency of moderate and severe VMS from baseline | Baseline to Weeks 1, 4, 8 and 12
  Frequency of moderate and severe VMS events will be calculated as the sum of moderate and severe VMS events per day. Percent reduction of >/= 75% will be reported.
Percent reduction at 100% in the frequency of moderate and severe VMS from baseline | Baseline to Weeks 1, 4, 8 and 12
  Frequency of moderate and severe VMS events will be calculated as the sum of moderate and severe VMS events per day. Percent reduction of 100% will be reported.
Pharmacokinetics (PK) of Fezolinetant in Plasma: Apparent Clearance (CL/F) for participants taking tamoxifen | Up to Week 24
  CL/F will be derived using a population PK model.
Pharmacokinetics (PK) of Fezolinetant in Plasma: Apparent Clearance (CL/F) for participants taking aromatase inhibitors | Up to Week 24
  CL/F will be derived using a population PK model.
PK of Fezolinetant in Plasma: apparent volume of distribution (Vc/F) for participants taking tamoxifen | Up to Week 24
  Vc/F will be derived using a population PK model.
PK of Fezolinetant in Plasma: apparent volume of distribution (Vc/F) for participants taking aromatase inhibitors | Up to Week 24
  Vc/F will be derived using a population PK model.
PK of Fezolinetant in Plasma: average concentration (Cavg) for participants taking tamoxifen | Up to Week 24
  Cavg will be derived using a population PK model.
PK of Fezolinetant in Plasma: Cavg for participants taking aromatase inhibitors | Up to Week 24
  Cavg will be derived using a population PK model.
PK of Fezolinetant in Plasma: trough concentration (Ctrough) for participants taking tamoxifen | Up to Week 24
  Ctrough will be derived using a population PK model.
PK of Fezolinetant in Plasma: Ctrough for participants taking aromatase inhibitors | Up to Week 24
  Ctrough will be derived using a population PK model.
PK of tamoxifen in Plasma: CL/F | Up to Week 24
  CL/F will be derived using a population PK model.
PK of tamoxifen in Plasma: Vc/F | Up to Week 24
  Vc/F will be derived using a population PK model.
PK of tamoxifen in Plasma: Cavg | Up to Week 24
  Cavg will be derived using a population PK model.
PK of tamoxifen in Plasma: Ctrough | Up to Week 24
  Ctrough will be derived using a population PK model.
PK of tamoxifen Metabolite 4-OH tamoxifen in Plasma: CL/F | Up to Week 24
  CL/F will be derived using a population PK model.
PK of tamoxifen Metabolite 4-OH tamoxifen in Plasma: Vc/F | Up to Week 24
  Vc/F will be derived using a population PK model.
PK of tamoxifen Metabolite 4-OH tamoxifen in Plasma: Cavg | Up to Week 24
  Cavg will be derived using a population PK model.
PK of tamoxifen Metabolite 4-OH tamoxifen in Plasma: Ctrough | Up to Week 24
  Ctrough will be derived using a population PK model.
PK of tamoxifen Metabolite N-desmethyltamoxifen in Plasma: CL/F | Up to Week 24
  CL/F will be derived using a population PK model.
PK of tamoxifen Metabolite N-desmethyltamoxifen in Plasma: Vc/F | Up to Week 24
  Vc/F will be derived using a population PK model.
PK of tamoxifen Metabolite N-desmethyltamoxifen in Plasma: Cavg | Up to Week 24
  Cavg will be derived using a population PK model.
PK of tamoxifen Metabolite N-desmethyltamoxifen in Plasma: Ctrough | Up to Week 24
  Ctrough will be derived using a population PK model.
PK of tamoxifen Metabolite endoxifen in Plasma: CL/F | Up to Week 24
  CL/F will be derived using a population PK model.
PK of tamoxifen Metabolite endoxifen in Plasma: Vc/F | Up to Week 24
  Vc/F will be derived using a population PK model.
PK of tamoxifen Metabolite endoxifen in Plasma: Cavg | Up to Week 24
  Cavg will be derived using a population PK model.
PK of tamoxifen Metabolite endoxifen in Plasma: Ctrough | Up to Week 24
  Ctrough will be derived using a population PK model.
PK of aromatase inhibitors in Plasma: CL/F | Up to Week 24
  CL/F will be derived using a population PK model.
PK of aromatase inhibitors in Plasma: Vc/F | Up to Week 24
  Vc/F will be derived using a population PK model.
PK of aromatase inhibitors in Plasma: Cavg | Up to Week 24
  Cavg will be derived using a population PK model.
PK of aromatase inhibitors in Plasma: Ctrough | Up to Week 24
  Ctrough will be derived using a population PK model.
Mean change from Baseline in the MENQOL Total Score | Baseline to Weeks 4, 8, 12 and 24
  The MENQOL is a 29-item PRO measure that assesses the impact of 4 domains of menopausal symptoms, as experienced over the last week: vasomotor, psychosocial, physical and sexual. The total score is the mean of the domain means. Higher scores represent more bothersome menopausal symptoms. A reduction (improvement) of 1 is the minimum clinically important difference for the MENQoL.
Mean change from Baseline in the MENQOL VMS 1-week recall domain score | Baseline to Weeks 4, 8 and 24
  The MENQOL is a 29-item PRO measure that assesses the impact of 4 domains of menopausal symptoms, as experienced over the last week: vasomotor, psychosocial, physical and sexual. Each item score ranges from 1 to 8, and each domain is scored separately; each domain mean ranges from 1 to 8. Higher scores represent more bothersome menopausal symptoms.
Mean change from Baseline in the MENQOL psychosocial 1-week recall domain score | Baseline to Weeks 4, 8, 12 and 24
  The MENQOL is a 29-item PRO measure that assesses the impact of 4 domains of menopausal symptoms, as experienced over the last week: vasomotor, psychosocial, physical and sexual. Each item score ranges from 1 to 8, and each domain is scored separately; each domain mean ranges from 1 to 8. Higher scores represent more bothersome menopausal symptoms.
Mean change from Baseline in the MENQOL physical 1-week recall domain score | Baseline to Weeks 4, 8, 12 and 24
  The MENQOL is a 29-item PRO measure that assesses the impact of 4 domains of menopausal symptoms, as experienced over the last week: vasomotor, psychosocial, physical and sexual. Each item score ranges from 1 to 8, and each domain is scored separately; each domain mean ranges from 1 to 8. Higher scores represent more bothersome menopausal symptoms.
Mean change from Baseline in the MENQOL sexual 1-week recall domain score | Baseline to Weeks 4, 8, 12 and 24
  The MENQOL is a 29-item PRO measure that assesses the impact of 4 domains of menopausal symptoms, as experienced over the last week: vasomotor, psychosocial, physical and sexual. Each item score ranges from 1 to 8, and each domain is scored separately; each domain mean ranges from 1 to 8. Higher scores represent more bothersome menopausal symptoms.
Mean change from Baseline in the PROMIS SD SF 8b Total (raw) Score | Baseline to Weeks 4, 8 and 24
  The PROMIS SD SF 8b assesses self reported sleep disturbance over the past 7 days and includes perceptions of: restless sleep; satisfaction with sleep; refreshing sleep; difficulties sleeping, getting to sleep or staying asleep; amount of sleep; and sleep quality. Responses to each of the 8 items range from 1 to 5 and the range of possible summed raw scores is 8 to 40. Higher scores on the PROMIS SD SF 8b indicate more of the concept measured (disturbed sleep).
Scores on the Patient Global Impression of Change (PGI-C) VMS | Up to Week 24
  The PGI-C VMS evaluates patient perceived change in hot flashes/night sweats from the initiation of treatment. Ratings range from (1) much better to (7) much worse.
Change from Baseline in the Patient Global Impression of Severity (PGI-S) VMS Score | Baseline to Weeks 4, 8, 12 and 24
  The PGI-S VMS evaluates patient perceived severity of hot flashes/night sweats. Ratings range from (1) no problems to (4) severe problems.
Scores on the PGI-C sleep disturbance (SD) | Up to Week 24
  PGI-C SD evaluates patient perceived change in sleep disturbance from the initiation of treatment. Ratings range from (1) much better to (7) much worse.
Change from Baseline in the PGI-S SD Score | Baseline to Weeks 4, 8, 12 and 24
  The PGI-S SD evaluates patient perceived severity of sleep disturbance. Ratings range from (1) no problems to (4) severe problems.
PGI-S SD response | Up to Week 24
  Proportion of patients achieving a response in PGI-S SD. The PGI-S SD evaluates patient perceived severity of sleep disturbance. Ratings range from (1) no problems to (4) severe problems. PGI-S SD response is defined as at least 2 levels of improvement on PGI-S SD from baseline. Non-response is defined as not achieving a response.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (115):
- Canada (9):
  - Site CA15019, Sarnia, Ontario
  - Site CA15016, Sault Ste. Marie, Ontario
  - Site CA15002, Montreal, Quebec
  - Site CA15001, Québec, Quebec
  - Site CA15004, Québec, Quebec
  - Site CA15003, Sherbrooke, Quebec
  - Site CA15020, Victoriaville, Quebec
  - Site CA15018, Barrie
  - Site CA15007, Trois-Rivières
- Czechia (11):
  - Site CZ42006, České Budějovice
  - Site CZ42003, Hořovice
  - Site CZ42002, Hradec Králové
  - Site CZ42011, Nový Jičín
  - Site CZ42001, Olomouc
  - Site CZ42005, Prague
  - Site CZ42008, Prague
  - Site CZ42013, Prague
  - Site CZ42004, Tábor
  - Site CZ42007, Vodňany
  - Site CZ42009, Vsetín
- Denmark (5):
  - Site DK45007, Aalborg
  - Site DE45003, Esbjerg
  - Site DK45009, Hillerød
  - Site DK45002, Næstved
  - Site DE45008, Sønderborg
- France (11):
  - Site FR33003, Angers
  - Site FR33001, Bayonne
  - Site FR33005, Bordeaux
  - Site FR33018, Bordeaux
  - Site FR33017, Caen
  - Site FR33016, Dijon
  - Site FR33013, Le Mans
  - Site FR33007, Lille
  - Site FR33012, Lyon
  - Site FR33008, Montpellier
  - Site FR33002, Saint-Herblain
- Germany (8):
  - Site GR49005, Essen, North Rhine-Westphalia
  - Site DE49001, Bottrop
  - Site DE49009, Leipzig
  - Site DE49007, Mönchengladbach
  - Site DE49010, München
  - Site GR49003, Münster
  - Site GR49011, Witten
  - Site GR49014, Wolfsburg
- Hungary (7):
  - Site HU36007, Budapest
  - Site HU36008, Budapest
  - Site HU36006, Debrecen
  - Site HU36001, Eger
  - Site HU36002, Kecskemét
  - Site HU36010, Salgótarján
  - Site HU36003, Székesfehérvár
- Italy (8):
  - Site IT39011, Bologna
  - Site IT39015, Genova
  - Site IT39003, Milan
  - Site IT39013, Mirano
  - Site IT39017, Pavia
  - Site IT39018, Reggio Emilia
  - Site IT39012, Terni
  - Site IT39014, Tricase
- Netherlands (8):
  - Site NL31014, Amsterdam
  - Site NL31010, Breda
  - Site NL31006, Dirksland
  - Site NL31001, Haarlem
  - Site NL31002, Rotterdam
  - Site NL31004, Rotterdam
  - Site NL31012, Rotterdam
  - Site NL31009, Terneuzen
- Poland (15):
  - Site PO48019, Poznan, Skorzewo
  - Site PO48005, Bialystok
  - Site PO48006, Bydgoszcz
  - Site PO48004, Katowice
  - Site PO48017, Katowice
  - Site PO48015, Krakow
  - Site PO48021, Krakow
  - Site PO48007, Lodz
  - Site PO48012, Lodz
  - Site PO48020, Piła
  - Site PO48002, Poznan
  - Site PO48018, Poznan
  - Site PO48010, Szczecin
  - Site PO48003, Świdnik
  - Site PO48001, Warsaw
- Spain (19):
  - Site ES34011, Barcelona
  - Site ES34020, Barcelona
  - Site ES34021, Barcelona
  - Site ES34010, Elche
  - Site ES34003, Girona
  - Site ES34005, Granada
  - Site ES34006, Jaén
  - Site ES34017, León
  - Site ES34007, Madrid
  - Site ES34019, Madrid
  - Site ES34022, Madrid
  - Site ES34023, Madrid
  - Site ES34015, Majadahonda
  - Site ES34002, Murcia
  - Site ES34014, Murcia
  - Site ES34008, Palma
  - Site ES34009, Seville
  - Site ES34024, Seville
  - Site ES34013, Valencia
- United Kingdom (14):
  - Site GB44008, Bebington, Birkenhead
  - Site GB44009, Guildford, Surrey
  - Site GB44018, Aberdeen
  - Site GB44019, Birmingham
  - Site GB44003, Bristol
  - Site GB44016, Cambridge
  - Site GB44006, Glasgow
  - Site GB44002, Liverpool
  - Site GB44020, Liverpool
  - Site GB44005, London
  - Site GB44017, Oxford
  - Site GB44001, Preston Lancashire
  - Site GB44012, Redhill
  - Site GB44010, Stroke on Trent

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Liao C, Pal L. Novel Pharmacotherapies for Menopausal Symptoms. Obstet Gynecol. 2025 Oct 1;146(4):473-486. doi: 10.1097/AOG.0000000000006025. Epub 2025 Aug 7. PMID 40773756